CLINICAL TRIAL: NCT03487900
Title: Is the Endoscopic Remission Evaluation, Using the CREDO 1 Index / Score in CD Patients in Clinical Remission at Baseline, Predictive of Sustained Clinical Remission Using a 2-year Follow up: a Multicenter Prospective Cohort Study
Brief Title: Is the Endoscopic Remission Evaluation, Using the CREDO 1 Index / Score in CD Patients in Clinical Remission at Baseline, Predictive of Sustained Clinical Remission Using a 2-year Follow up
Acronym: CREDO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: AbbVie (Industry); Biogen (Industry); Celgene (Industry); Gilead Sciences (Industry); Roche Pharma AG (Industry); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GETAID 2017-002; 2017-003345-15 (EudraCT Number)
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: CD
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical remission CD (Other)
  Interventions: Diagnostic Test: Colonoscopy

INTERVENTIONS:
Diagnostic Test: Colonoscopy — Colonoscopy for CD patients in clinical remission

SUMMARY:
The CREDO 2 study follows CREDO 1 study, which aims to construct an objective evaluation of endoscopic remission in Crohn's Disease (CD). In addition to reproducibility and validation, the predictive value of this remission evaluation needs to be tested in different settings to valorise its usefulness in clinical practice and in clinical trials.

CREDO 2 aims to investigate whether the evaluation of endoscopic remission, as defined in CREDO 1, in patients in clinical remission is predictive of sustained clinical remission at 2 years.

The design of CREDO2 is a multicentre longitudinal prospective cohort study. The screening period to include a patient is two weeks. Patients will be followed up to week 104.

DETAILED DESCRIPTION:
The CREDO 2 study follows CREDO 1 study, which aims to construct an objective evaluation of endoscopic remission in Crohn's Disease (CD). In addition to reproducibility and validation, the predictive value of this remission evaluation needs to be tested in different settings to valorise its usefulness in clinical practice and in clinical trials.

CREDO 2 aims to investigate whether the evaluation of endoscopic remission, as defined in CREDO 1, in patients in clinical remission is predictive of sustained clinical remission at 2 years. The design of CREDO2 is a multicentre longitudinal prospective cohort study. The screening period to include a patient is two weeks. Patients will be followed up to week 104. The primary endpoint is sustained clinical remission at week 104. The primary secondary endpoints are sustained clinical remission at weeks 26 and 52. The sustained clinical remission at 2 years is defined by the absence of relapse and complication of the disease. Relapse is defined as Crohn's Disease Activity Index (CDAI) > 220 or between 150 and 220 for 2 consecutive weeks with an increase of at least 70 points relative to the baseline CDAI, associated with an objective marker of inflammation: C-reactive protein (CRP) ≥5 mg/l and / or faecal calprotectin ≥250 μg/g. CD complication is defined by an intestinal resection surgery for CD, stricturoplasty, endoscopic dilatation, hospitalisation for intestinal strictures, abscess and / or fistula (including anoperineal disease) and/or therapeutic escalation. Therapeutic escalation is defined as an increase in the dosage of the treatment, shortening of the treatment interval, addition of a new treatment for CD (including corticosteroids, immunosuppressants, biologics, Janus kinase (JAK) inhibitors or any experimental treatment). The number of patients to be included is 320 when using a two-sided test with a type 1 error of 5% to detect with a power of 80% an association between a predictor and week 104 sustained remission failure, corresponding to a variation in proportions of patients who failed from 40% in the high-risk group to 20% in the low-risk group, and assuming a 12% loss due to treatment discontinuation or patient withdrawal. Patients will be recruited via two cohorts. First, patients included in CREDO 1 could be included in CREDO 2 if they agree and meet the criteria of non-exclusion. Assuming that 2/3 of the 15 patients included in each of the 16 centres involved in CREDO 1 could be included in CREDO 2, 160 patients will be included from CREDO 1. An additional cohort of 10 patients per centre will be included in CREDO 2 by the same local investigator within each centre using the same methods as for CREDO 1 cohort, except that recruitment criteria will be those of CREDO 2, to provide 160 additional patients to reach the targeted cohort size for CREDO 2. Recruitment will therefore be performed in 16 centres and each local investigator will have to register 20 videos, including those selected from CREDO 1, stratified by endoscopic remission status according to his/her global judgment: complete remission; almost complete remission; neither complete nor almost complete remission. The main inclusion criteria are adult patients, with established CD with ileal and / or colonic involvement, without significant clinical activity for more than 3 consecutive months with, at baseline, CDAI <150 and CRP <5 mg / l and faecal calprotectin <250 μg / g, stable maintenance treatment for more than 3 months, an ileocolonoscopy planned for CD and the decision to maintain or decrease the treatment (but not increase) after the colonoscopy. All maintenance treatments are authorized / immunosuppressive (azathioprine, 6-mercaptopurine, methotrexate), biologic (infliximab, adalimumab, certolizumab, golimumab, ustekinumab, vedolizumab) and JAK inhibitors.The main exclusion criteria are an incomplete record of the ileocolonoscopy or more than three resected ileocolonic segments (not counting ileocecal valve), taking NSAIDs in the two weeks prior to endoscopy, anoperineal MC without luminal involvement, suspicion of intestinal infection within 4 weeks prior to baseline endoscopic assessment. The expected period of recruitment is 12 months from the first patient included in the study and 20 patients will be included in each of the 16 centres in Belgium and France. At inclusion, demographic, phenotypic, medical history and treatment data will be collected and ileocolonoscopy will be performed and recorded by the local investigator using pre-specified standards, provided sufficient quality. Biological (albumin, haemoglobin, platelets, CRP and faecal calprotectin) assessments will be carried out at the inclusion and at each follow-up visit (week 26, 52 104 and unplanned). The clinical activity will be evaluated through CDAI. Within each centre, the local investigator, as local reader, will read the 20 ileocolonoscopy videos of the centre. In addition, each video will be read by central readers, selected among 12 central readers in four groups of 3 central readers. Each video will be read by 2 central readers and by a third one in case of disagreement between the first two. Each central reader will read a little more than 54 videos due to these disagreements. All these readers, local and central, will have undergone the training session validated by an examination on the evaluation of endoscopic remission. In a separate delayed session, the central readers will evaluate components of usual endoscopic severity indices. Agreement between data provided by local readers and central readers will be assessed through Kappa and intraclass correlation coefficient estimates. If agreement is satisfactory, endoscopic data provided by local readers will be used to investigate the association between baseline endoscopic evaluation and sustained clinical remission at week 104 using the logistic regression method, ROC curves, sensitivity and specificity. If agreement is poor, the association will be studied on central reader data using the same methods.

This study should provide a tool to evaluate the ability of endoscopic remission evaluation in patients in clinical remission to accurately predict sustained clinical remission. If it is the case, this tool could become the therapeutic objective for patients in clinical remission with ileal and/or colonic CD. If agreement is satisfactory between local and central reading, the tool could be used in therapeutic trials, but also in clinical practice. If this is not the case, the tool should be used in clinical trials using central readings.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 year of age
2. Established CD for more than 6 months with histopathological confirmation available in the medical records of the patient
3. Clinical remission as considered by the investigators global assessment ≥3 consecutive months
4. Clinical remission at baseline (CDAI <150) and CRP <5 mg/l and fecal calprotectin <250 μg/g
5. CD maintenance treatment needs to be stable for ≥3 months before baseline
6. Planned ileocolonoscopy for CD
7. Permitted maintenance treatment for CD: immunomodulators (Azathioprine, 6-mercaptopurine, methotrexate), biologicals (infliximab, adalimumab, certolizumab, golimumab, ustekinumab, vedolizumab) and JAK inhibitors
8. No planned escalation of treatment after baseline endoscopy
9. The subject signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures

Exclusion Criteria:

1. Pregnancy at time of endoscopy
2. People unable to give their consent (because of their physical or mental state).
3. Absence of written consent.
4. Ulcerative colitis or IBD type unclassified
5. Specific postsurgical settings: ileoanal anastomosis, ileostomy or colostomy
6. Incomplete recording of the endoscopy or more than three resected ileocolonic segments (not counting ileocecal valve)
7. Non-steroidal anti-inflammatory drugs intake within two weeks before baseline endoscopy
8. Perianal fistulizing CD without luminal disease
9. Contraindication for endoscopy
10. Inaccessible ileocolonic segment even after attempt of endoscopic balloon dilation
11. Suspicion of gastrointestinal infection within 4 weeks prior to baseline endoscopy
12. Documented active or suspicion of intestinal tuberculosis
13. Conditions which in the opinion of the investigator may interfere with the subject's ability to comply to the follow up with the study procedures.

    CREDO2-GT2017002 Getaid_CREDO2-Protocol_v1.1_20171130 Page 18 of 37
14. Exclusive CD of the upper gastrointestinal tract (Montreal classification L4)
15. Montreal classification L1 without terminal ileal involvement
16. Colon preparation with solutions other than PEG or picosulphate solutions
17. Incomplete recording of the baseline endoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained clinical remission at week 104 | Week 104

SECONDARY OUTCOMES:
Sustained clinical remission at week 52 | Week 52
Sustained clinical remission at week 26 | Week 26
Time to disease flare based on biomarker measurement | Week 104
Sustained clinical remission according to treatment group as an exploratory endpoint | Week 104

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (4):
  - AZ Sint Lucas Gent, Ghent
  - Leuven University Hospital, Leuven
  - UZ Leuven, Leuven
  - CHU Liège, Liège
- France (10):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU Estaing - Clermont Ferrand, Clermont-Ferrand
  - APHP- Hopital BEAUJON, Clichy
  - CHRU de Lille - Hôpital C. Huriez, Lille
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - CHU Nancy - Hôpital Barbois, Nancy
  - CHU Nantes - Hôtel Dieu, Nantes
  - CHU de Nice - Hôpital de l'Archet 2, Nice
  - Hôpital Saint Antoine, Paris
  - CHU Bordeaux - Hôpital Haut Lévêque, Pessac

IPD SHARING:
Plan to Share IPD: Undecided
ND